CLINICAL TRIAL: NCT02259530
Title: Sustainable and Adapted Treatment Strategies to Restore Psychological Functioning and Mental Health Among Displaced Somalis: Preparation of a Multicenter Treatment Study (P114/02/2014): Pilot Study 3.
Brief Title: Case Series for Traumatized Refugees With Khat Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: Africa Institute of Mental and Brain Health (AFRIMEB) (Other)
Responsible Party: Principal Investigator, Michael Odenwald, Researcher, University of Konstanz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01DG13020_a
Record Dates: First submitted 2014-09-30; First posted 2014-10-08 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Posttraumatic Stress Disorder; Khat Use Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Integrated Psychotherapeutic Intervention (Experimental): Integrated treatment of khat use disorder and PTSD
  Interventions: Behavioral: Integrated Psychotherapeutic Intervention

INTERVENTIONS:
Behavioral: Integrated Psychotherapeutic Intervention — Evidence-based standard tools for the treatment of PTSD and comorbid khat dependence: Community Reinforcement Approach, Relapse Prevention, Narrative Exposure Therapy

SUMMARY:
The research project will offer psychotherapeutic treatment to Somali refugees with PTSD and comorbid khat dependence. In this case series, evidence-based techniques will be applied and adapted to the cultural background of Somali refugees in Kenya.

DETAILED DESCRIPTION:
More than 500.000 Somali refugees live in Kenya. This group is especially burdened by high rates of exposure to traumatic events, high prevalence of PTSD and a high comorbidity with substance use disorders, mainly related to khat (catha edulis). There's a shortage of literature on psychotherapeutic methods that are applicable in this group. The aim of this case series is to develop modifications of standard therapeutic techniques to the Somali culture and to the needs of this group. Twenty successive cases will be recruited from a community clinic where refugees often seek for treatment because of psychiatric problems. Senior level psychotherapists will apply and adapt techniques and approaches like Community Reinforcement Approach (CRA), Relapse Prevention (RP), and Narrative Exposure Therapy (NET); all sessions will be video recorded. Regular supervision with external experts and group discussions will be held to evaluate and adapt the single procedures and techniques. The aim of this study is the development of a standardized approach that can be used in a Randomized Controlled Trial which will be conduced in the future.

ELIGIBILITY:
Inclusion Criteria:

PTSD (DSM-IV) Khat Dependence (DSM-IV)

Exclusion Criteria:

Severe Psychotic Disorder Suicidality Mental Disability

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Posttraumatic Stress Diagnostic Scale (PDS) | 3 months
  Pre-post change of self-reported PTSD-symptom severity
Time-Line Follow Back(TLFB) | 3 months
  Pre-post change of self-reported days with khat use

SECONDARY OUTCOMES:
Hopkins Symptom Checklist (HSCL) | 3 months
  Pre-post change of self-reported depressive symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Africa Mental Health Foundation, Nairobi, Kenya